CLINICAL TRIAL: NCT02702050
Title: A Prospective Randomized Clinical Trial to Investigate the Effect of Mechanical Stimulation on Mastectomy Scars
Brief Title: Effect of Mechanical Stimulation on Mastectomy Scars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Queen Elizabeth Hospital (Other)
Responsible Party: Principal Investigator, Ka Po Andrea LEUNG, Senior Physiotherapist, The Queen Elizabeth Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KC/KE-15-0816/FR-3
Record Dates: First submitted 2016-02-26; First posted 2016-03-08 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: Physiotherapy; Mechanical Stimulation; Mastectomy Scar
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional treatment group (Active Comparator): Conventional treatment group will receive an educational session before commencement of the program. Twelve sessions of 40-minute remedial exercises, 5-minute warm up and 5-minute cool down exercises will be provided within a 6-week period (i.e., two sessions per week) to all subjects. No mechanical stimulation will be given.
  Interventions: Other: Conventional treatment
- Mechanical stimulation group (Experimental): A 10 minute mechanical stimulation program - 'Mechanical stimulation (LPG system; Cellu M6 Integral I), will be provided after each of the twelve sessions of conventional treatment.
  Interventions: Other: Mechanical stimulation (LPG system; Cellu M6 Integral I)

INTERVENTIONS:
Other: Mechanical stimulation (LPG system; Cellu M6 Integral I) — For the mechanical stimulation group, an additional ten-minute mechanical stimulation will be provided in each of the twelve sessions of convention treatment program. The device produced skin lift through suction via a treatment head with 2 rollers installed. It was a non-invasive technique which aimed to mobilize soft tissues by creating skin folds and stretching the underlying soft tissues while manipulating the treatment head according to protocol.
  Other Names: Therapeutic massager
  Arms: Mechanical stimulation group
Other: Conventional treatment — Twelve sessions of 40-minute remedial exercises, 5-minute warm up and 5-minute cool down exercises, within a 6-week period (i.e., two sessions per week)
  Arms: Conventional treatment group

SUMMARY:
The purpose of this study is to investigate the efficacy of mechanical stimulation on mastectomy scars in:

(i) alleviating scar appearance - pigmentation, vascularity, pliability and thickness, (ii) reducing shoulder morbidities, (iii) improving arm functions, and (iv) enhancing quality of life, in women with breast cancer after mastectomy.

DETAILED DESCRIPTION:
Background:

Breast cancer is common among women. After surgical interventions like mastectomies, women with breast cancer may suffer physical, emotional and psychosocial complications. Evidence suggests that comprehensive physiotherapy program, including patient education, manual techniques, therapeutic exercises and compression bandaging, is effective in managing the above complications. Scarring was frequently overlooked in past studies. Besides cosmetic issues, a post mastectomy scar may cause adverse physical, functional, and psychological outcomes. The effects of mechanical stimulation on mastectomy scars have not been well investigated yet.

Objectives:

To investigate the efficacy of mechanical stimulation in:

(i) alleviating scar appearance - pigmentation, vascularity, pliability and thickness, (ii) reducing shoulder morbidities, (iii) improving arm functions, and (iv) enhancing quality of life, in women with breast cancer after mastectomy.

Setting:

Out-patient physiotherapy breast care clinic at the Hong Kong Queen Elizabeth Hospital

Participants:

One hundred and eight women with breast cancer after mastectomy in recent 6 weeks will be recruited.

Methodology:

An assessor-blind, randomized controlled trial will be conducted. 108 women with breast cancer after mastectomy will be recruited from the breast care clinic of the Queen Elizabeth Hospital. They will be randomly allocated by block randomization method into either the mechanical stimulation group (n= 54) or conventional treatment group (n=54).

Both study groups will receive an educational session before commencement of the program. Twelve sessions of 40-minute remedial exercises, 5-minute warm up and 5-minute cool down exercises will be provided within a 6-week period (i.e., two sessions per week) to all subjects. For the mechanical stimulation group, a ten-minute mechanical stimulation program will be provided. For the conventional treatment group, no mechanical stimulation will be given.

Primary outcomes include scar evaluations by the Vancouver Scar Scale and spectrophotometry. Secondary outcomes are composite measurements of shoulder morbidities, including numeric pain rating scale (NPS), shoulder range of movement and hand grip strength; arm function as evaluated by the Disabilities of the Arm, Shoulder and Hand (DASH-HKPWH) questionnaire; and quality of life as measured by the Functional Assessment of Chronic Illness Therapy - Breast Cancer (FACT-B). Outcome assessments at baseline, immediately after the 6-week program, and 3-month follow-up periods will be conducted by blinded assessors at the breast care clinic.

Data Analysis:

The results will be analyzed using two-way repeated measures analysis of variance with Statistical Package for Social Sciences version 21.0. Alpha level will be set at 0.05.

Potential Clinical Significance of Study:

Improvement of physiotherapy in scar management might potentially improve scar appearance - pigmentation, vascularity, pliability and thickness, decrease shoulder morbidities, improve upper limb functions, and enhance quality of life for women with breast cancer after mastectomy. If the mechanical stimulation protocol is proven to be effective, it will bring about significant advances in physiotherapy practice in post-mastectomy care in an evidence-based manner.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years old or above with mastectomy performed in recent 6 weeks;
* Able to attend physiotherapy treatment and follow-ups during the study period.

Exclusion Criteria:

* Altered mental state for cooperation and informed consent;
* Signs and symptoms of mastectomy scar infections or inflammations;
* Unhealed mastectomy wounds;
* History of lymphoedema;
* Diagnosed bilateral breast cancers;
* Unstable medical or cardiovascular conditions;
* Pre-existing arm impairments/dysfunctions that will affect testing or exercising the affected arm;
* Receiving radiotherapy during the study period;
* Known sensitivity to mechanical stimulation;
* Skin cancer on the treatment area;
* Unclear cut margins of the cancer;
* Known metastasis to other areas;
* HIV positive.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Vancouver Scare Scale (VSS) to study scar appearance | 6 months
  A scar scale to quantify scar appearance by observing the thickness, pliability, pigmentation and vascularity of mastectomy scar. The former two items were rated on ordical scales whereas the later two items in a descriptive manner. Total score ranged from 0 to 13.
Spectrophotometry to measure scar color | 6 months
  A spectrophotometer (Hunterlab Miniscan Ez4500S, USA) is used to measure level of lightness, redness and yellowness of the mastectomy scar versus adjacent normal skin. Level of redness indicated vascularization and pigmentation represented significance of melanin deposited in a scar.

SECONDARY OUTCOMES:
Numeric pain rating scale (NPS) to study pain over affected breast | 6 months
  11-item numeric rating scale (NRS) is valid, reliable and appropriate for use in clinical setting for pain measurement
Shoulder range by goniometry | 6 months
  Shoulder range of motion (ROM) will be evaluated by measuring active shoulder flexion and abduction
Grip strength by hand-held dynamometer | 6 months
  The hand grip strength will be evaluated using the JAMAR Hydraulic Hand Dynamometer
Arm function | 6 months
  The Chinese version of the Disabilities of the Arm, Shoulder and Hand (DASH-HKPWH) questionnaire will be used as an outcome measurement for upper extremities disabilities and symptoms.
Quality of life | 6 months
  The Functional Assessment of Chronic Illness Therapy - Breast Cancer (FACT-B), traditional Chinese version 4 questionnaire would be adopted for measurement of quality of life for women with breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Andrea KP LEUNG, MSc, Principal Investigator — Physiotherapy Department ,Queen Elizabeth Hospital
Locations (1):
- Queen Elizabeth Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No